CLINICAL TRIAL: NCT00524017
Title: Phase II Study of Single-Agent Cetuximab for Treatment of High-Risk Pre-malignant Upper Aerodigestive Lesions
Brief Title: Cetuximab in Treating Patients With Precancerous Lesions of the Upper Aerodigestive Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J0644 CDR0000562250; P50CA096784 (NIH); P30CA006973 (NIH); JHOC-J0644; JHOC-NA_00001757
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Cancer; Precancerous Condition
Keywords: hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; precancerous condition
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (treatment) (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, and 50 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab
- Arm II (control) (No Intervention): Patients receive regular follow-up care

INTERVENTIONS:
Biological: cetuximab — given IV
  Arms: Arm I (treatment)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block abnormal cell growth in different ways. Some block the ability of abnormal cells to grow and spread. Others find abnormal cells and help kill them or carry cell-killing substances to them.

PURPOSE: This randomized phase II trial is studying how well cetuximab works in treating patients with precancerous lesions of the upper aerodigestive tract.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the histologic response rate in patients with high-risk, premalignant lesions of the upper aerodigestive tract treated with cetuximab.

Secondary

* To determine the clinical response rate in these patients.
* To determine if patterns of epidermal growth factor receptor (EGFR) component expression are altered in these patients.
* To determine the change in status of genetic alterations, including loss of heterozygosity, in these patients.

OUTLINE: This is a multicenter study. Patients are stratified by lesion type [diffuse dysplasia vs recurrent dysplasia vs dysplastic lesions with 3p or 9p loss of heterozygosity (LOH)]. Patients are randomized to 1 of 2 arms.

* Arm I (treatment): Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, and 50 in the absence of disease progression or unacceptable toxicity.
* Arm II (control): Patients receive regular follow-up care. Patients have the option of receiving cetuximab after completion of the study.

In both arms, patients with persistent or recurrent high-grade dysplasia or dysplastic lesions with 3p or 9p LOH undergo surgical resection, if feasible, after week 8.

Tumor biopsy samples are obtained at baseline* and after week 8 for histologic and biomarker correlative studies. Tissue samples are analyzed by histopathology to determine histologic changes in post-treatment lesions and by immuno-histochemistry (IHC) to measure expression and activation of EGFR signaling pathway components. LOH studies are also performed.

NOTE: *Paraffin-embedded tissue from the original diagnostic biopsy may be used for baseline assessment, if the diagnostic biopsy was performed within 3 months prior to study entry.

After completion of study therapy, patients are followed at approximately 1 month, every 3 months for 2 years, and then every 6 months for up to 5 years as per routine standard of care.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk, premalignant lesions of the upper aerodigestive tract, meeting one of the following criteria:

  * Unresectable, diffuse high-grade dysplasia, defined as moderate or severe dysplasia that is not assessable by physical examination and/or that cannot be excised by standard surgical techniques
  * previously treated HNSCC with persistent or recurrent high grade dysplasia with no evidence of head and neck malignancy for three months prior to enrollment or who have successfully completed therapy for head and neck malignancy more than 3 months prior to enrollment.
  * Dysplastic lesions with 3p or 9p loss of heterozygosity
* Disease location amenable to endoscopic biopsy in an outpatient clinical setting or operative biopsy within the routine scheduling and practice of clinical care

  * No medical contraindication to biopsy of the target lesion
  * Pathology must be reviewed by the Johns Hopkins Hospital Department of Pathology

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) > 1,000/mm³
* Platelet count > 75,000/mm³
* Creatinine clearance > 60 mL/min
* Total serum bilirubin < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No concurrent illness likely to preclude study therapy or surgical resection
* Patients with a history of a curatively treated malignancy are eligible provided they are disease-free and have a survival prognosis that exceeds 5 years
* No evidence of clinically active interstitial lung disease

  * Patients with chronic, stable radiographic changes who are asymptomatic are eligible
* No history or radiological evidence of pulmonary fibrosis
* No acute myocardial infarction within the past 3 months
* No uncontrolled angina, arrhythmia, or congestive heart failure
* No evidence of other severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No evidence of any other significant clinical disorder or laboratory finding that would preclude study participation
* No known severe hypersensitivity to cetuximab or any of its excipients
* No prior hypersensitivity reaction to chimerized or murine monoclonal antibody therapy
* No severe abnormality of the cornea

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior oncologic or other major surgery or biopsy
* More than 30 days since prior non-approved or investigational drugs
* No prior chemotherapy, radiotherapy, or surgery for the premalignant lesions
* No prior EGFR-targeted agents (e.g., cetuximab, gefitinib, or erlotinib)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Califano, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (10):
- United States (9):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled patients with premalignant lesions of the Head and Neck with mild, moderate or severe dysplasias
Pre-assignment Details: 16 participants did not have biopsy proven dysplasia as required by protocol and were not randomized to treatment.
Period: Overall Study
Arm/Group | Arm I (Treatment) | Arm II (Control)
Started | 13 | 6
Completed | 13 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Treatment) | Arm II (Control) | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 7 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Based on Histologic Grade
Description: Histologic downgrade by at least one grade of dysplasia (e.g Severe to Moderate).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 13 | 6
Participants | 13 | 6

2. Secondary Outcome: Number of Participants With Objective Response Based on Clinical Assessment
Description: Clinical visualization on whether lesion responded to treatment (i.e., direct visualization of the lesion combined with histologic grade)
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 13 | 6
Participants | 13 | 6

3. Secondary Outcome: Status of Epidermal Growth Factor Receptor (EGFR) Pathway Components and Molecular Alterations in Pre-treatment Biopsies
Time Frame: Baseline (pre-treatment)
Population: Data was not collected for this outcome
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Status of EGFR Pathway Components and Molecular Alterations in Post-treatment Biopsies
Time Frame: At 8 weeks post-treatment
Population: Data was not collected for this outcome
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Survival
Time Frame: Up to year 5 years post-treatment
Population: No patients were followed for this outcome measure
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Lesion Recurrence
Time Frame: Up to year 5 years post-treatment
Population: No patients were followed for this outcome measure
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Treatment) | Arm II (Control)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 0/13 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No